CLINICAL TRIAL: NCT00363662
Title: Diagnostic Utility of MRI in Intracerebral Hemorrhage
Acronym: DASH
Status: Completed | Type: Observational
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Marion S Buckwalter, Principle Investigator, Stanford University
Other Study IDs: 2R01NS034866-08A1 (NIH)
Record Dates: First submitted 2006-08-09; First posted 2006-08-15 (Estimated); Last update posted 2021-11-17 (Actual); Status verified 2021-11

CONDITIONS: Cerebral Hemorrhage
MeSH Terms: conditions — Cerebral Hemorrhage

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

SUMMARY:
The overall aim of this project is to prospectively determine whether MRI can improve the conventional neuroradiological evaluation (CT with or without cerebral angiography) of patients with a spontaneous ICH or IVH. The study design will also allow us to identify the added benefit of specific MR sequences and repeat MRI in the chronic stage, thereby allowing us to prospectively determine their value in a consecutive series of patients. This information should have a major impact on the management of these patients by providing data on the diagnostic yield of routine MRI in patients presenting with a wide variety of causes for ICH or IVH. These data will help guide the diagnostic evaluation and the management of brain hemorrhage patients in the future.

DETAILED DESCRIPTION:
Spontaneous intracerebral hemorrhage (ICH) and intraventricular hemorrhage (IVH) account for at least 15% of strokes worldwide. There are many possible etiologies for spontaneous (i.e. non-traumatic) ICH or IVH such as longstanding hypertension and cerebral amyloid angiopathy.

Other causes include vascular malformations, intracranial aneurysms, tumors, coagulopathies, use of thrombolytic or antithrombotic drugs, cerebral venous thrombosis, hemorrhagic transformation of an ischemic infarct, illicit drug use, endocarditis, and vasculitis.

Identification of the cause of an ICH or IVH typically relies on clinical evaluation supported by computer tomography (CT) with or without conventional contrast cerebral angiography in selected patients. While magnetic resonance imaging (MRI) has substantially improved our diagnostic capabilities, the appropriate use of MRI and its effectiveness has not been studied systematically in these patients. Furthermore, it is unclear whether routine MRI in ICH yields clinically relevant data. For this reason routine use or MRI in patients with ICH is highly variable in clinical practice. Furthermore, it is unclear whether the findings detected on MRI will change management decisions regarding further diagnostic testing and therapeutic options above and beyond that which can be achieved by CT and cerebral angiography.

This question has major ramifications for the care of patients with ICH or IVH. If MRI truly can categorize patients into specific diagnostic categories better than CT, this would represent a major paradigm shift in the way that these patients are typically evaluated. On the other hand, because of the added expense of MRI, its general use could result in a substantial increase in the cost of neurological care. These added costs must result in improvements in patient management in order to justify the added financial resources involved.

The overall aim of this project is to prospectively determine whether MRI can improve the conventional neuroradiological evaluation (CT with or without cerebral angiography) of patients with a spontaneous ICH or IVH. The study design will also allow us to identify the added benefit of specific MR sequences and repeat MRI in the chronic stage, thereby allowing us to prospectively determine their value in a consecutive series of patients. This information should have a major impact on the management of these patients by providing data on the diagnostic yield of routine MRI in patients presenting with a wide variety of causes for ICH or IVH. These data will help guide the diagnostic evaluation and the management of brain hemorrhage patients in the future. During this 5-year study, 160 consecutive inpatients presenting with a spontaneous ICH or IVH within 48 hours of symptom onset will be prospectively categorized into specific hemorrhage subtypes based upon the findings on MRI. We will:

1. Prospectively assess the value of early MRI in determining hemorrhage etiology in consecutive patients who present with a spontaneous ICH or IVH diagnosed by CT. We will test the hypotheses that:

   1. MRI will more frequently yield a correct specific hemorrhage etiology than conventional non-contrast CT.
   2. MRI will increase the certainty of a specific hemorrhage etiology when compared to conventional non-contrast CT.
   3. MRI will affect management in patients who present with a spontaneous ICH or IVH diagnosed by CT.
   4. The yield of MRI in patients with a spontaneous ICH or IVH varies among diagnostic categories.
   5. Routine use of MRI in patients with spontaneous ICH or IVH will reduce the need for conventional (and invasive) cerebral angiography in these patients.
2. Prospectively assess the relative added value of an improved MR protocol (MRA/MRV, GRE, DWI, TEDS, PROPELLER) in the evaluation and management of patients with ICH or IVH determined by non-contrast CT.

   We will test the hypotheses that:

   a. MRI with multi-echo, multi-shot GRE sequences, MRA, MR venography (MRV), SENSE-DWI and PROPELLER-DWI will more accurately assign patients into appropriate diagnostic categories than conventional MRI (T1W, T1W post gadolinium, T2W [FSE/FLAIR FSE]) and CT.
3. Prospectively identify the added benefit of repeated MRI in the chronic stage in the evaluation and management of patients with ICH or IVH. We will test the hypotheses that:

   1. Repeat MRI in the chronic stage (at 60 days) will yield a specific ICH etiology above and beyond early MRI and CT.

This information will contribute substantially to our understanding of the value of routine MRI in patients with a spontaneous ICH or IVH both in the acute and in the chronic phase. It will also allow us to develop practice guidelines for the use of MRI in these patients.

ELIGIBILITY:
Inclusion Criteria:

A. Men and non-pregnant women, at least 18 years of age.

B. Patients with an ICH or IVH admitted to Stanford University Medical center within 48 hours of symptom onset.

C. Ability to undergo MRI.

Exclusion Criteria:

A. Patients with a known (preexisting) source for ICH, for example a known untreated arterio-venous malformation.

B. Patients receiving investigational drug therapies or procedures prior to MRI scanning.

C. Glasgow coma scale (GCS) score < 6 in the absence of sedating medications.

D. Informed consent cannot be obtained either directly from the patient or from a legally authorized representative.

E. Severe coexisting or terminal systemic disease that limits life expectancy or that may interfere with the conduct of the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: A total of 180 ICH or IVH patients will be studied. All patients will be inpatients admitted to the Stanford Stroke Center, a multidisciplinary referral center for the treatment of acute stroke. Consecutive patients will be enrolled provided they meet the inclusion and exclusion criteria and that they or a legally authorized representative give informed consent.
Sampling Method: Probability Sample
Enrollment: 180 (Actual)
Dates: Start 2006-06-26 (Actual); Primary Completion 2010-01-27 (Actual); Study Completion 2010-01-27 (Actual)

PRIMARY OUTCOMES:
Diagnostic comparison | Approximately 60 minutes to acquire each scan.
  Compare the diagnosis by the treating physician (based on the patient history, examination, CT, and angiography results) with the treating physician's diagnosis based on additional review of the MRI. The CT-based diagnosis and the MRI-based diagnosis by the treating physician will be compared to the "gold standard" diagnosis reached by the outside adjudication panel (which excludes information from the MRI studies).

CONTACTS AND LOCATIONS:
Overall Officials: Gregory Albers, MD, Principal Investigator — Stanford University
Locations (1):
- Stanford University School of Medicine, Stanford, California, United States